CLINICAL TRIAL: NCT01849367
Title: Trial of Bilateral tDCS for Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC13052
Record Dates: First submitted 2013-05-05; First posted 2013-05-08 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tDCS (1) (Experimental)
  Interventions: Device: Eldith Neuroconn tDCS device
- Active tDCS (2) (Active Comparator)
  Interventions: Device: Eldith Neuroconn tDCS device

INTERVENTIONS:
Device: Eldith Neuroconn tDCS device

SUMMARY:
Transcranial direct current stimulation (tDCS) is a novel treatment approach for depression that has shown promising efficacy in four recent double-blind, randomized, sham-controlled trials (RCT) and a meta-analysis. Mood, cognitive test performance and biomarkers will be measured during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Participant meets criteria for a DSM-IV Major Depressive episode.
2. MADRS score of 20 or more.

Exclusion Criteria:

1. Diagnosis (as defined by DSM-IV) of: any psychotic disorder (lifetime); eating disorder (current or within the past year); obsessive compulsive disorder (lifetime); post-traumatic stress disorder (current or within the past year); mental retardation.
2. History of drug or alcohol abuse or dependence (as per DSM-IV criteria) within the last 3 months (except nicotine and caffeine).
3. Inadequate response to ECT in the current episode of depression.
4. Participant is on regular benzodiazepine medication which is not clinically appropriate to discontinue.
5. Participant requires a rapid clinical response due to inanition, psychosis or high suicide risk.
6. Neurological disorder or insult, e.g., recent stroke (CVA), which places participant at risk of seizure or neuronal damage with tDCS.
7. Participant has metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
8. Female participant who is pregnant, or of child-bearing age, sexually active and not using reliable contraception (urine test for pregnancy will be used).
9. Participants who are not fluent in English will not be included in the trial for safety reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 4 weeks

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Black Dog Institute / University of New South Wales, Sydney, New South Wales, Australia